CLINICAL TRIAL: NCT03415919
Title: Collection of Gastrointestinal Malignant and Non-malignant Human Samples
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Hyun Jung Kim, Assistant Professor, University of Texas at Austin
Other Study IDs: IRB 2017-06-0114
Record Dates: First submitted 2018-01-16; First posted 2018-01-30 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Inflammatory Bowel Diseases; Colo-rectal Cancer
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood, diseased tissue, normal tissue, and fecal matter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IBD patients: Patients suffering from IBD scheduled to have a biopsy by colonoscopy.
  Interventions: Other: no intervention will be given to patients.
- CRC patients: Patients suffering from CRC scheduled to have a biopsy by colonoscopy, or surgical resection of colon.
  Interventions: Other: no intervention will be given to patients.
- Control patients: Patients who are scheduled to have a colonoscopy for routine screening to serve as a control population.

INTERVENTIONS:
Other: no intervention will be given to patients. — samples are collected at the time of a scheduled procedure that is part of normal treatment. This study will not have any impact on the care or treatment the patient receives.
  Groups: CRC patients; IBD patients

SUMMARY:
To collect human tissue, blood, and fecal samples from patients suffering from Inflammatory Bowel Disease and Colorectal Cancer. The samples will be used to establish biomimetic human organ-on-a-chip technology, as well as study the role of the microbiome in the pathogenesis in human gastrointestinal diseases.

DETAILED DESCRIPTION:
The purpose of the proposed research is to collect tissue, blood and fecal samples from patients undergoing standard of care for their gastrointestinal disease, including Inflammatory Bowel Disease (IBD), and Colorectal Cancer (CRC). Tissue and blood samples will be obtained during procedures that are part of normal treatment, including blood and fecal collection, surgical resection, and biopsy collection. Samples will be obtained from consenting patients at Seton Dell Medical Center at the University of Texas (SDMCUT), or other relevant facilities (see section 6.i below), and only tissue not required for histopathological analysis will be collected. Initially, the focus will be on IBD, and CRC, where there are extensive previous studies to draw from.

The collected samples of the proposed study will be used to establish biomimetic human organ-on-a-chip platforms by leveraging microfluidic tissue culture technology. Another focus of the research will be study the human intestinal microbiome that is highly associated with the pathogenesis of human gastrointestinal diseases. The investigators have developed the microchip technology to mimic the structure and physiological function of human intestine by integrating tools developed in a microfluidic device, tissue engineering, and clinical microbiology, using intestinal cell lines. To recreate more reliable intestinal disease models and to further investigate the host-gut microbiome interactions in these experimental platforms, the investigators are transitioning to use human clinical samples. The investigators will use tissue biopsies to culture human intestinal cells including epithelium, endothelium, connective tissues on-chip. Blood samples will also obtained to isolate peripheral blood mononuclear cells (PBMC) that represent mixed population of white blood cells (WBC). Isolated WBCs will be co-cultured with intestinal cells. Any potential application of microbiome-related therapies such as fecal microbiota transplantation (FMT) will also be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven colorectal cancer scheduled to have surgical resection of primary site, at participating and approved facilities. Since it is standard clinical care to resect certain suspicious gastrointestinal masses without a pre-existing biopsy, patients who are undergoing resections for highly suspicious masses believed to be cancer, may be consented.
* Diagnosed with Inflammatory Bowel Disease (IBD) or Crohn's Disease (CD), scheduled to have biopsy and/or fecal collection.
* scheduled to have a colonoscopy as part of routine screening.

  * 18 years old.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* The study will not exclude potential subjects from participation on the basis of ethnic origin or gender. Subjects recruited will include men, women, and all ethnic origins, provided they meet all inclusion criteria listed above.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No special populations are targeted for accrual to this study. However, racial background may play a role in disease etiology, and a variety of races is optimal for this study to address that question. Thus, the patient's race information will be included with the sample.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-07-13 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
confirmation of diagnosis by pathologist | directly following procedure
  Once tissue is collected, those samples that have a confirmed diagnosis of disease by the pathologist will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jung Kim, PhD, Principal Investigator — Assistant Professor; Richard D Fleming, MD, FACS, Principal Investigator — Associate Director for Surgical Services
Locations (1):
- The University of Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
no protected health information will be shared with other researchers. Experimental data, and samples obtained during this study may be shared with other researchers.

DOCUMENTS (1):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03415919/Prot_001.pdf